CLINICAL TRIAL: NCT03521466
Title: A Randomized Control Trial Evaluating the Effectiveness of a Medical Student Guided Smoking Cessation Program for Hospitalized Smokers in India
Brief Title: Medical Student Counseling for Hospitalized Patients Addicted to Tobacco
Acronym: MS-CHAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Government Calicut Medical College (Unknown); Wayanad Institute of Medical Sciences (Unknown); PSG Institute of Medical Science and Research (Other)
Responsible Party: Principal Investigator, Richard Josephson, MS MD, Director CVP Rehabilitation, Harrington Heart and Vascular Institute, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 01-18-11
Record Dates: First submitted 2018-04-14; First posted 2018-05-11 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Smoking Cessation Counselling; Medical Student Education
Keywords: Smoking cessation counselling; Medical Student education; India

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Coordinators calling the patient to assess quit status are blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Smoking Cessation counseling by trained medical students with or without Nicotine Replacement Therapy
  Interventions: Behavioral: Smoking Cessation Counseling
- Control (No Intervention): The control group will receive counseling and/or NRT at the discretion of the treating physician.

INTERVENTIONS:
Behavioral: Smoking Cessation Counseling — Trained medical students will visit patients inpatient while hospitalized and provide smoking cessation counseling and recommend Nicotine Replacement Therapy. They will continue to follow these patients for 2 months after discharge and provide telephone-based counseling.
  Arms: Intervention

SUMMARY:
The purpose of this randomized control trial is two- fold. The primary hypothesis of the study is that smoking cessation counseling delivered through trained medical students will lead to higher rates of abstinence amongst patients in the intervention group, as compared to a control group, when measured by self-reported and biochemical testing at 6 months after enrolment .

The secondary hypothesis is that medical students engaging in a structured curriculum that includes counseling hospitalized smokers will show demonstrable increases in knowledge, confidence in their abilities, and use of smoking cessation techniques in regular practice.

DETAILED DESCRIPTION:
India is the 2nd largest consumer of tobacco in the world, with 275 million Indians using tobacco. Each hospitalization is an opportunity for providers to motivate their patients to quit. However, the Indian medical curriculum typically offers little training in the skills required to successfully counsel a patient to quit smoking. The investigators hypothesize that trained medical students can increase subsequent quit rates among hospitalized smokers, while acquiring skills in tobacco cessation counseling.

The investigators propose a 2-armed multicenter randomized controlled trial (RCT) that will compare the effectiveness of standard hospital practice versus a medical student-guided smoking cessation program initiated inpatient and continued for three months after discharge. The target study population includes current smokers admitted to the general medicine, pulmonary and cardiology wards. These patients will be randomized to receive either usual care or the intervention. The intervention group will receive both inpatient and longitudinal post-discharge telephone counseling by medical students who have successfully completed a training workshop in tobacco cessation counseling and pharmacotherapy. The students can also recommend nicotine replacement therapy (NRT) to the patient if indicated. The control group will receive counseling and/or NRT at the discretion of the treating physician. They will not receive phone based counseling after discharge.

Patients from both groups will be asked to report their quit status 6 months after enrolment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 18-70 years old, who are admitted to the medical, and if required surgical wards.
2. Patients must be current smokers (cigarettes and/or bidis) at the time of admission or report having smoked at all in the last 4 weeks prior to admission (to account for changes in behaviour during illness).
3. Patients living within 10 Km radius of the hospital.

Exclusion Criteria:

1. Unwilling to participate
2. Patients who use only non-smoked tobacco will be excluded.
3. Patients who are are daily alcohol users, daily cannabis or psychotropic drug users.
4. Patients who do not have a telephone/ unable to follow up
5. Patients unable to understand the local/common language
6. Patients with psychiatric conditions rendering them incapable of interacting with the providers
7. Medically unstable patients
8. Patients with expected hospital stay <24 hours
9. Patients with life expectancy < 12 months
10. Pregnant patients
11. Patients currently participating in a tobacco cessation program
12. Prior participation in this trial during another hospitalisation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
Biochemically verified 7 day quit rate measured 6 months after enrolment. | 6 months from enrolment
  At 6 months from enrolment, patients will be asked to report abstinence from smoking over the last 7 days (No more than 5 cigarettes in total since quit date); those who claim to have quit will be asked to provide biochemical confirmation by exhaled carbon monoxide breath testing (<10 Parts Per Million will be considered a verified quit attempt).

SECONDARY OUTCOMES:
Biochemically verified 90 day quit rate, measured 6 months after enrolment | 6 months from enrolment
  At 6 months from enrolment, patients will be asked to report abstinence from smoking over the last 90 days; those who claim to have quit will be asked to provide confirmation by exhaled carbon monoxide breath testing (<10 Parts Per Million will be considered a verified quit attempt)
Number of patients achieving a 50% reduction in the number of cigarettes /bidis smoked in a week, measured at 2 and 6 months after enrolment | 2 and 6 months from enrolment
Correlation between verified quit rates at 6 months and FTND scores at enrolment | 6 months from enrolment
Number of patients who report having quit smoking in the last 7 days (irrespective of biochemical verification) | 2 and 6 months from enrolment
Agreement between self reported quit 7 day quit rate and biochemically verified 7 day quit rate, measured at 6 months from enrolment | 6 months from enrolment
No of patients who have refrained from using smokeless tobacco in the last 7 days, measured at 6 months. | 6 months from enrolment
Pre-post analysis of medical student knowledge about counseling techniques and pharmacotherapy | 6 weeks and 12 months after training
  Students will be given a knowledge questionnaire before training and 6 weeks after training. The questionnaire will be scored from 0 to 22, 0 being the lowest and 22 being the highest score.
Qualitative analysis of student attitudes towards smoking cessation counseling | 12 months after training
  Assessed by surveying students who participated in counseling patients. Some questions will be scored on a Likert scale ranging from 1-5; Others are open ended questions and will be analyzed to identify relevant themes.
Qualitative analysis of the feasibility and acceptability of the intervention | 12 months after training
  Students who participate in the trial will receive a survey with open ended questions. The responses will be analysed to identify relevant themes.

OTHER OUTCOMES:
Number of eligible patients that receive inpatient counseling and atleast 3 follow up calls | 2 months from enrolment
  Data from the patient screening and follow up forms will be used to calculate this ratio
Number of patients who use any form of cessation pharmacotherapy within the first 2 months | 2 months from enrolment
  Patients will be asked to report the use of pharmacotherapy during their 2 month follow up call
Number of patients enrolled in the study that are available for follow up at 6 months | 6 months from enrolment

CONTACTS AND LOCATIONS:
Locations (1):
- PSG Institute of Medical Science and Research, Coimbatore, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Satish P, Khetan A, Shah D, Srinivasan S, Balakrishnan R, Padmanandan A, Hejjaji V, Hull L, Samuel R, Josephson R. Effectiveness of Medical Student Counseling for Hospitalized Patients Addicted to Tobacco (MS-CHAT): a Randomized Controlled Trial. J Gen Intern Med. 2023 Nov;38(14):3162-3170. doi: 10.1007/s11606-023-08243-y. Epub 2023 Jun 7. PMID 37286774